CLINICAL TRIAL: NCT04911452
Title: Creating a CALMER NICU: Pilot Testing a Robot for Optimizing Growth and Brain Development in Preterm Infants in the NICU
Brief Title: Creating a Calmer NICU: Optimizing Growth and Brain Development in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Women's Health Research Institute of British Columbia (Other)
Responsible Party: Principal Investigator, Manon Ranger, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H21-00527
Record Dates: First submitted 2021-05-22; First posted 2021-06-03 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Prematurity
Keywords: Prematurity; Neonatal intensive care; Growth; Robotic device; Skin-to-skin care; Stress; Brain activity; EEG
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Single-site, single-blind, two-group (treatment and control), randomized pilot trial
Who Masked: Outcomes Assessor
Masking Description: Data outcomes for growth and clinical data will be blind to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard Neonatal Intensive Care Unit (NICU) care
- Calmer (Experimental): Calmer placed and left in infant incubator for a minimum of 2 and maximum of 3 weeks.
  Calmer treatment provided for minimum total of 3 hours/day (can be discontinuous).
  Interventions: Device: Calmer

INTERVENTIONS:
Device: Calmer — Once randomized, infants in the Calmer group will receive treatment for a minimum cumulative total of 3 hours/day during periods when the infant may be too ill to be held or when parents do not wish to hold their infant or are not present. Calmer does not replicate a parent's contact and so the minimum exposure has been tripled. No upper limit of Calmer use will be set. Each day, the research and/or bedside nurse will record the heart and respiratory rates for a two-minute period. The one-minute average will be used to program Calmer for each infant that day to better simulate day-to-day changes in infant-parent contact. The Neonatal Intensive Care Unit (NICU) research nurse will also train the parents/caregivers to self-measure their resting heart and breathing rates so that if they are away from the NICU for more than one day, these values can be sent to the research/ bedside nurse by phone.
  Arms: Calmer

SUMMARY:
Infants born preterm can spend months in the neonatal intensive care unit (NICU) where they experience stressful but essential procedures. Untreated stress is associated with altered brain development. Skin-to-skin care (SSC) is one of the most effective behavioral strategies for mitigating preterm infant stress and improving brain maturation. However, parents may not be always available to provide SSC; some infants cannot be held for long periods for medical reasons. To address this problem, investigators designed Calmer, a patented, prototype therapy bed, for reducing stress in preterm infants. Calmer fits into NICU incubators and provides simultaneously an artificial skin surface, heartbeat sounds and breathing motion, mimicking aspects of SSC; the latter 2 features are individualized for each infant based on their parents' recordings. The 1st randomized controlled trial (RCT) in 58 preterm babies showed that during a routine blood test: Calmer lowered infant behavioral and heart stress responses and stabilized brain blood flow no differently than facilitated tucking; infants could be cared for safely on Calmer up to 6 hours in 1 day; Calmer was well accepted by mothers and staff.

The goal now is to determine the efficacy of Calmer use over 3 weeks to support optimal physical growth and brain development in preterm infants. A 2-group (treatment, control) pilot RCT to test the implementation of an increased "dose" of Calmer exposure over 2-3 continuous weeks is proposed. 30 infants born between 26-30 weeks gestational age in the NICU will be randomized to receive either Calmer, for a minimum of 3 hours in total/day for 2-3 continuous weeks, or to 2-3 weeks of standard NICU care (minimum of 2 and maximum of 3 weeks).

Research questions:

Trial feasibility Q1. Is it feasible to enrol 30 infants, complete a 2-3-week treatment period (minimum of 2 and maximum of 3 weeks), and measure growth outcomes in preterm infants (26-30 weeks GA) in the NICU in a pilot RCT of daily Calmer treatment versus standard NICU care to inform a larger, definitive RCT?

Infant outcomes Q2a. Are there differences in physical growth markers (daily weight gain, head circumference, body length) between preterm infants who receive Calmer and those who receive standard NICU care measured before (baseline) and after 2-3 weeks of daily Calmer exposure? Q2b. Are there differences in brain activity markers, as measured by cerebral electrical (EEG) signalling, between preterm infants who receive Calmer and those who receive standard NICU care, measured during a resting/sleeping state and routine diaper change session at the end of the trial (post 2-3 weeks of daily Calmer exposure)?

DETAILED DESCRIPTION:
Pilot trial implementation targets:

Targets for success would be that the informed consent rate will be at least 40%, 30 patients will be enrolled in 48 months, 95% of infants will receive the 3 hour minimum treatment, and patient assessment completion rate will be at least 85%.

The results of this pilot trial will be used to inform the design of a larger RCT. The results of this pilot trial will allow to assess patient accrual, protocol adherence, and to monitor the completeness and quality of the outcome data. If implementation targets are met, an application for further funding to use this protocol in a larger, multisite, non-inferiority trial comparing SSC + Calmer to SSC alone will be put forth.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants admitted to the neonatal intensive care unit (NICU) at the British Columbia (BC) Women's Hospital born at 26-30 completed weeks gestational age (GA). GA is determined accurately using early gestation ultrasonogram (standard of care in BC), or calculated using the last menstrual period;
* Infants who are on continuous positive airway pressure or are ventilated;
* At least one parent/caregiver must speak sufficient English to provide consent

Exclusion Criteria:

* Infants who have congenital anomalies, small for GA (per medical admission history), or have a history of maternal abuse of controlled drugs and substances; - Infants with an ongoing infection at the time of enrolment;
* Infants that have pre-existing cardiovascular instability defined by shock/hypotension/need for cardiovascular drugs
* Infants receiving paralytic drugs;
* Infants that have major neurological injury (e.g. hypoxic ischemic encephalopathy, hemorrhage/stroke);
* Infants who are beyond the 30th completed week GA (30 weeks + 6 days) at enrolment.

Ages: 26 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Trial feasibility: Consent rates | 48 months
  Overall average consent rate of infants/month
Trial feasibility: Protocol delivery rate | 48 months
  Percent of on/off protocol infants for the trial period
Trial feasibility: Complete outcome measures | 48 months
  Percent of infants with complete clinical primary and secondary outcome measures
Trial feasibility: Safety issues | 48 months
  Rate of safety issues identified

SECONDARY OUTCOMES:
Brain activity at rest and during stress event (routine diaper change) | 2-3 weeks
  EEG measure during a single session (at end of the 3-week). EEG assessments for ~60 min when the infants are at rest in their incubator (undisturbed during quiet/active sleep) while laying on the Calmer device turned off (if experimental group, otherwise incubator as standard).
  EEG measurements will be taken in 4 phases:
  1. Baseline A: 15-minute Sleep + Calmer device OFF (Pre)
  2. Baseline B: 15-minute Sleep + Calmer device ON
  3. Stressful event: Diaper change (standardized) + Calmer device ON
  4. Recovery: 15-minute Sleep + Calmer device ON
  We will conduct brain activity EEG measurements using a 64-channel HydroCel Geodesic Sensor Net specifically designed to suit the very small heads and fragile skin of preterm infants (EGI, Eugene, OR). We will have synchronized bedside video recordings and code stress behaviours using the NICU standard pain assessment tool.
Weight gain | 2-3 weeks
  The change in average infant weight gain between Calmer and control groups in grams/day (g/d) will be measured on the day before the start of the treatment (baseline), at the mid-way point (~day 11), and at the end of the 3-week period, then divided by the number of treatment days. Sex and gestational age (GA) age-specific percentiles for the measures will be calculated using the Fenton Growth charts. Changes in weight percentiles between baseline and end of treatment will then be calculated.
Nutritional status | 2-3 weeks
  Measures of daily feeding and nutritional data will include: method of feeding (intravenous, nasogastric, oral-gastric, oral), type (total parenteral nutrition, breastmilk (mother's or donor), formula, additives (Human milk fortifier, lipids), frequency/timing and method (breast/bottle) of transition from tube to oral feeds at transfer/discharge.
Head circumference | 2-3 weeks
  Baseline, mid-point and end-of-treatment measures of head circumference in cm (occipito-frontal circumference [OCP]) will be reported. Sex and GA age-specific percentiles for the measures will be calculated using the Fenton Growth charts. Changes in OFC percentiles between baseline and end of treatment will then be calculated.
Body length | 2-3 weeks
  Baseline, mid-point and end-of-treatment measures of body length in cm will be reported. Sex and GA age-specific percentiles for the measures will be calculated using the Fenton Growth charts. Changes in body length percentiles between baseline and end of treatment wil then be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Holsti, PhD, Principal Investigator — The University of British Columbia; Manon Ranger, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- British Columbia Women's Hospital and Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnston C, Campbell-Yeo M, Disher T, Benoit B, Fernandes A, Streiner D, Inglis D, Zee R. Skin-to-skin care for procedural pain in neonates. Cochrane Database Syst Rev. 2017 Feb 16;2(2):CD008435. doi: 10.1002/14651858.CD008435.pub3. PMID 28205208
- [Background] Holsti L, MacLean K, Oberlander T, Synnes A, Brant R. Calmer: a robot for managing acute pain effectively in preterm infants in the neonatal intensive care unit. Pain Rep. 2019 Mar 14;4(2):e727. doi: 10.1097/PR9.0000000000000727. eCollection 2019 Mar-Apr. PMID 31041426
- [Background] Ranger M, Albert A, MacLean K, Holsti L. Cerebral hemodynamic response to a therapeutic bed for procedural pain management in preterm infants in the NICU: a randomized controlled trial. Pain Rep. 2021 Jan 12;6(1):e890. doi: 10.1097/PR9.0000000000000890. eCollection 2021 Jan-Feb. PMID 33490850
- [Background] Williams N, MacLean K, Guan L, Collet JP, Holsti L. Pilot Testing a Robot for Reducing Pain in Hospitalized Preterm Infants. OTJR (Thorofare N J). 2019 Apr;39(2):108-115. doi: 10.1177/1539449218825436. Epub 2019 Feb 15. PMID 30770034
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Background] Hauser S, Suto MJ, Holsti L, Ranger M, MacLean KE. Designing and Evaluating Calmer, a Device for Simulating Maternal Skin-to-Skin Holding for Premature Infants. In Proceedings of the 2020 CHI Conference on Human Factors in Computing Systems (CHI '20). 2020. Association for Computing Machinery, New York, NY, USA: 1-15. https://doi.org/10.1145/3313831.3376539